CLINICAL TRIAL: NCT07155304
Title: Percutaneous Sigmoid Fixation For Management Of Recurrent Sigmoid Volvulus : A Randomized Controlled Trial
Brief Title: Percutaneous Sigmoid Fixation For Management Of Recurrent Sigmoid Volvulus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Said Mohamed Said Abdou Negm, assistant professor of general surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mahmoud Alballat
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Endoscopic Surgical Procedure
Keywords: endoscopy, volvulus,
MeSH Terms: conditions — Intestinal Volvulus

STUDY DESIGN:
Intervention Model Description: The investigators included all patients who were presented to emergency department with recurrent sigmoid volvulus at Zagazig University hospital between (August 2024 to August 2025). Sample size in this study was calculated based on comparison of mortality rate after endoscopy and surgical procedure in elderly patients with sigmoid volvulus as primary outcome for this study. Prior data from (Jackson et al., 2020) revealed that mortality rate after surgical intervention was 16-42% and after percutaneous fixation was 9.7%. So, using power and sample size calculator we included 33 patients in the surgical group(group1) and 33 patients in the percutaneous group (group2) to be able to reject the null hypothesis that mortality rates for both groups' subjects were equal with probability (power) 0.8. The type I error probability associated with this test of this null hypothesis was 0.05. We used an uncorrected chi-squared statistic to evaluate this null hypothesis. Dropout rate was 20%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- percutaneous group (Active Comparator): percutaneous fixation of sigmoid volvulus after endoscopic untwisting to prevent recurrence using anchor device
  Interventions: Procedure: percutaneous sigmoid colon fixation
- surgical group (No Intervention): surgical management of sigmoid volvulus

INTERVENTIONS:
Procedure: percutaneous sigmoid colon fixation — after endoscopic sigmoid colon untwisting , percutaneous colon fixation using anchor device
  Arms: percutaneous group

SUMMARY:
The investigators included all patients who were presented to emergency department with recurrent sigmoid volvulus at Zagazig University hospital between (August 2024 to August 2025). The investigators included patients were of the American Society of Anesthesiologists (ASA) Physical status I-II-III-IV, high risk surgical patients and patients with age of 16-80 years old while excluded patients with ASA V, VI, patients with lower abdominal surgery and obese patients with body mass index more than 35. This prospective randomized controlled clinical trial was approved by Zagazig University Faculty of Medicine Institutional Review Board (Approval Number: 633/1-Sep-2024) and performed in accordance with the code of ethics of the World Medical Association (Declaration of Helsinki) for studies involving human subjects.

DETAILED DESCRIPTION:
The investigators included all patients who were presented to emergency department with recurrent sigmoid volvulus at Zagazig University hospital between (August 2024 to August 2025). The investigators included patients were of the American Society of Anesthesiologists (ASA) Physical status I-II-III-IV, high risk surgical patients and patients with age of 16-80 years old while excluded patients with ASA V, VI, patients with lower abdominal surgery and obese patients with body mass index more than 35. This prospective randomized controlled clinical trial was approved by Zagazig University Faculty of Medicine Institutional Review Board (Approval Number: 633/1-Sep-2024) and performed in accordance with the code of ethics of the World Medical Association (Declaration of Helsinki) for studies involving human subjects.

Sample size in this study was calculated based on comparison of mortality rate after endoscopy and surgical procedure in elderly patients with sigmoid volvulus as primary outcome for this study. Prior data from (Jackson et al., 2020) revealed that mortality rate after surgical intervention was 16-42% and after percutaneous fixation was 9.7%. So, using power and sample size calculator we included 33 patients in the surgical group and 33 patients in the percutaneous group to be able to reject the null hypothesis that mortality rates for both groups' subjects were equal with probability (power) 0.8. The type I error probability associated with this test of this null hypothesis was 0.05. We used an uncorrected chi-squared statistic to evaluate this null hypothesis. Dropout rate was 20%.

Primary outcome was recurrence of the sigmoid volvulus while the secondary outcomes were mortality rate , complications and hospital stay in each group after the intervention during the 3-months follow-up period, respectively.

Follow up after endoscopy and discharge from the hospital All patients were clinically examined, and laboratory checked during the hospital stay. Any suspected gastric leak post repair mandated CT scan with oral and I.V contrast and upper GI endoscopy. After discharge, patients who had undergone balloon dilation as a part of their repair procedure were scoped every 4 weeks to continue the dilation till relief of distal pouch narrowing. Patients were followed-up for at least 3 months post repair.

Statistical analysis Analysis of data was performed using SPSS (Statistical Package of Social Services) version 22. Quantitative variables were described as mean (±SD, standard deviation) and median (range) according to Shapiro test of normality. Qualitative variables were described as number and percentage. Chi-square test was used to compare qualitative variables between the 2 groups. Fisher exact test was used when one expected cell or more are less than 5. Unpaired t-test was used to compare quantitative variables, in parametric data (SD < 30% of the mean). Mann Whitney test was used instead of unpaired t-test in non-parametric data (SD > 30% of the mean). The results were considered statistically significant when the significant probability was less than 0.05 (P < 0.05). P-value < 0.001 was considered highly statistically significant (HS), and P-value ≥ 0.05 was considered statistically insignificant (NS).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical status I-II-III-IV, high risk surgical patients and patients with age of 16-80 years old

Exclusion Criteria:

* patients with ASA V, VI, patients with lower abdominal surgery and obese patients with body mass index more than 35

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
incidence of recurrence of volvulus | within one week after the endoscopy
  incidence of recurrence of volvulus

CONTACTS AND LOCATIONS:
Overall Officials: Said Mohamed Negm, M.D, Principal Investigator — Zagazig University Faculty Medicine
Locations (1):
- Zagazig University, Zagazig, Sharquia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided